CLINICAL TRIAL: NCT02781519
Title: Gender Related Differences in the Acute Effects of Delta-9-Tetrahydrocannabinol in Healthy Humans
Acronym: THC-Gender
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1505015940
Record Dates: First submitted 2016-05-16; First posted 2016-05-24 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- THC (Active Comparator): Active THC (0.015mg/kg) administered intravenously over 10 minutes.
  Interventions: Drug: THC
- Placebo (Placebo Comparator): Control: small amount of alcohol intravenously (quarter teaspoon), with no THC over 10 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC — Active THC (0.015mg/kg) administered over 10 minutes
  Other Names: Delta-9-Tetrahydrocannabinol
  Arms: THC
Drug: Placebo — Control: small amount of alcohol (quarter teaspoon), with no THC over 10 minutes
  Arms: Placebo

SUMMARY:
The purpose of the study is to characterize the acute effects of cannabinoids in women relative to men and to begin probing the mechanisms that may underlie gender differences.

ELIGIBILITY:
Inclusion Criteria:

* at least one lifetime exposure to cannabis
* good physical and mental health

Exclusion Criteria:

* cannabis naive individuals
* major current or recent stressors
* taking estrogen supplements or oral contraceptive pills (for women)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rewarding Effects measured by Visual Analog Scale (VAS) | changes in "high" assessed over the following timepoints: baseline, +10, +80, and +200 minutes after THC infusion begins
  subjective measure of THC induced "high"
Verbal Learning: measured by Rey Auditory Verbal Learning Test (AVLT) | 25 minutes after THC infusion begins
  measured as delay recall on the AVLT

CONTACTS AND LOCATIONS:
Locations (1):
- Biological Studies Unit at the VA Connecticut Healthcare System, Yale School of Medicine, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohammad Aghaei A, Urban Spillane L, Pittman B, Flynn LT, De Aquino JP, Bassir Nia A, Ranganathan M. Sex differences in the acute effects of oral THC: a randomized, placebo-controlled, crossover human laboratory study. Psychopharmacology (Berl). 2024 Oct;241(10):2145-2155. doi: 10.1007/s00213-024-06625-6. Epub 2024 Jun 4. PMID 38832949